CLINICAL TRIAL: NCT07223021
Title: Improving EveNt Free Survival by Optimizing FLUdarabine Exposure During LymphodepletioN for CAR T CEll Therapy: a Randomized, Multi-center Study of Children and Young Adults With B-cell Acute Lymphoblastic Leukemia (INFLUENCE)
Brief Title: A Study of Fludarabine Dosing in Children and Young Adults With B-cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Princess Maxima Center for Pediatric Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-072
Record Dates: First submitted 2025-10-28; First posted 2025-10-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: Fludarabine
MeSH Terms: conditions — Burkitt Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: The study is a randomized open-label multicenter trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Fludarabine regimen followed by CAR-T (Active Comparator): Fludarabine 30 mg/m2/dose x 4 doses on days -6 to -3 (or -7 to -4)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CAR-T
- Targeted fludarabine regimen followed by CAR-T (Experimental): Fludarabine 40 mg/m2/dose x 2 doses on days -6 and -5 (or -7 and -6), with doses on days -4 and -3 (or -5 and -4, if starting lymphodepletion on day -7) adjusted based on PK analysis to target a cumulative area under the curve (AUC) of 18 mg*h/L (range 17.5-18.5mg*h/L
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: CAR-T

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2/dose x 4 doses on days -6 to -3 (or -7 to -4)
  Arms: Standard Fludarabine regimen followed by CAR-T
Drug: Cyclophosphamide — All patients will receive Cyclophosphamide 500 mg/m2 IV on days -6 and -5 (or -7 and -6).
Drug: Fludarabine — Targeted fludarabine LD: Fludarabine 40 mg/m2/dose x 2 doses on days -6 and -5 (or
  -7 and -6), with doses on days -4 and -3 (or -5 and -4, if starting lymphodepletion on day -7) adjusted based on PK analysis to target a cumulative area under the curve (AUC) of 18 mg*h/L (range 17.5-18.5mg*h/L)
  Arms: Targeted fludarabine regimen followed by CAR-T
Biological: CAR-T — will be infused based on institutional guidelines.

SUMMARY:
The researchers are doing this study to find out whether PK-targeted fludarabine is an effective Lymphodepletion (LD) chemotherapy approach for people with relapsed/refractory B-cell acute lymphoblastic leukemia (B-ALL) who will receive tisagenlecleucel CAR T-cell therapy. The researchers will compare PK-targeted fludarabine dosing with standard fludarabine dosing to see which treatment approach is more effective. The researchers will also look at whether PK-targeted fludarabine dosing is feasible (practical), the side effects of the study treatment, and how the study treatment affects people's quality of life. The researchers will measure quality of life by having participants complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-ALL and eligible to receive commercial tisagenlecleucel.
* Patient's weight > 9 kg at time of lymphodepleting chemotherapy
* Adequate organ function at time of LD is required and is defined:

  * Hepatic: Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia
  * Hepatic: AST and ALT < 5x the upper limit of normal for age, unless thought to be leukemic disease-related
  * Renal: Calculated glomerular filtration rate (GFR) ≥ 70 ml/min/1.73m^2. (based on Schwartz formula GFR (mL/min/1.73 m²) = (36.2 × Height in cm) / Creatinine in μmol/L
  * Cardiac: LVEF ≥ 50% by multi-gated acquisition scan (MUGA), resting echocardiogram, or cardiac magnetic resonance imaging (MRI) within 6 weeks of screening
  * Pulmonary: Oxygen saturation as recorded by pulse oximetry of ≥ 90% on room air
* Adequate performance status:

  * Age ≥ 16 years: ECOG ≤ 1 or Karnofsky > 60% at treatment
  * Age < 16 years: Lansky ≥ 60% at treatment
* Willing to participate as research subject and provide written informed consent from parents/legal representative, patient, and age-appropriate assent as appropriate before any study specific screening procedures are conducted, according to local, regional or national law and legislation.

Exclusion Criteria:

* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to the study drugs, or drugs chemically related to study treatment or excipients that contraindicate their participation, including fludarabine, cyclophosphamide and tisagenlecleucel.
* Patients with tisagenlecleucel that is deemed out of specification (OOS) will be excluded from this protocol
* Clinically significant active and uncontrolled infection confirmed by clinical evidence, imaging, or positive laboratory tests (e.g., blood cultures, PCR for DNA/RNA etc.)
* Patient/parent/guardian unable to give informed consent or unable to comply with the treatment protocol.
* Pregnant or lactating women

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
compare the event free survival (EFS ) | 28 days
  EFS is defined as time from randomization until non-response at day 28 after CAR T cell infusion, loss of B-cell aplasia <6 months from the time of CAR T cell infusion, disease relapse, initiation of anti-leukemic therapy or death of any cause

SECONDARY OUTCOMES:
survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Curran, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/